CLINICAL TRIAL: NCT01277952
Title: Deep Brain Stimulation for Treatment of Severe Disability From Traumatic Brain Injury
Brief Title: Deep Brain Stimulation for Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai, MD (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, MD, MD, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2010H0264
Record Dates: First submitted 2011-01-13; First posted 2011-01-17 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; DBS
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DBS Surgery (Experimental): Deep brain stimulation (DBS) will be the treatment option in this study along with behavioral interventions for participants with severe disability due to Traumatic Brain Injury (TBI) 24 months post their injury, the participants will have severe disabilities in behavioral and emotional self-regulation, cognitive impairments and somatic symptoms.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Brain pace maker, implanted in the brain
  Other Names: DBS

SUMMARY:
The study will evaluate the benefit of Deep Brain Stimulation for subjects with severe disability due to Traumatic Brain Injury.

DETAILED DESCRIPTION:
The study will evaluate the benefit of Deep Brain Stimulation for subjects with severe disability due to Traumatic Brain Injury. DBS has been proven safe and efficacious for remediation of multiple neurological conditions. It is the hope of the study team that the protocol will provide further insight into the potential of DBS to improve the quality of life and functioning of persons with severe disability due to TBI and at the same time can provide new clinical insights that will improve treatment for the entire spectrum of injury severity.

ELIGIBILITY:
Inclusion Criteria:

* 24 months post traumatic brain injury Scores in Severe range of the Glasgow Outcome Scale-Extended Evidence of impaired cognitive functioning Medically and neurologically stable

Exclusion Criteria:

* Medical contraindications for surgery Evidence of substance abuse in the last 12 months Current Diagnosis of major depressive disorder current participation in rehabilitation services Co-morbid conditions that would interfere with study activities

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Improvement in Brain Functioning | 16 months
  Brain functioning improvement in functional independence, community participation and subjective well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No